CLINICAL TRIAL: NCT06617338
Title: Native Alignment in the Setting of an Arthritic Knee in Total Knee Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Arthur Malkani, Orthopedic Surgeon, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 24.0701
Record Dates: First submitted 2024-09-25; First posted 2024-09-27 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-01

CONDITIONS: Osteoarthritis (OA) of the Knee
Keywords: osteoarthritis; knee; total knee arthroplasty; target alignment
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Prospective, randomized cohort analysis study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Participant receives bilateral knee CT preoperatively (Experimental): The P.I. (Dr. Malkani) will use normal contralateral side joint numbers as the target alignment for RA-TKA
  Interventions: Diagnostic Test: CT scan bilateral knee
- Participant receives unilateral CT of the operative knee preoperatively (Active Comparator): The P.I. will use the traditional method to obtain target alignment for RA-TKA.
  Interventions: Diagnostic Test: CT scan unilateral knee

INTERVENTIONS:
Diagnostic Test: CT scan unilateral knee — Intervention given to the Active Comparator arm
  Arms: Participant receives unilateral CT of the operative knee preoperatively
Diagnostic Test: CT scan bilateral knee — Intervention given to the Experimental Arm
  Arms: Participant receives bilateral knee CT preoperatively

SUMMARY:
The goal of this clinical trial is to learn if preparing the target alignment of the operative side in total knee arthroplasty (TKA) based on the non-arthritic side will give the patient better overall alignment, function, and improved results compared to basing our implant alignment and positioning off the arthritic side, which is currently the traditional method.

The main questions it aims to answer are:

* Will a patient have improved postoperative TKA results if the implant alignment is based off the non-arthritic side compared to the standard arthritic side?
* What are the similarities or differences between study arms with respect to final implant alignment and positioning angles? Researchers will compare the outcomes of two cohorts of patients undergoing primary robotic-assisted total knee arthroplasty (RA-TKA) with normal contralateral knee. Based on preoperative CT imaging, the researchers will use normal contralateral side joint numbers as the target alignment for one group (Experimental arm) and utilize the traditional method for the other group (Active comparator arm). Clinical outcomes and patient-reported outcome measures (PROMs) will be compared between groups.

Participants will:

* Be randomized into one of two study arms and will receive either a unilateral knee CT or bilateral knee CT preoperatively
* Follow-up in the clinic at 2 weeks, 6 weeks and 1-year postoperatively, per standard-of-care for x-ray and clinical evaluation.
* Complete postop questionnaires (PROMs) at the prescribed follow-up intervals

ELIGIBILITY:
Inclusion Criteria:

1. Patient age is 21-89 at time of surgery
2. Patient is indicated to undergo a unilateral primary TKA, secondary to osteoarthritis
3. Patient's contralateral knee is non-arthritic
4. Patient agrees to participate as a study subject and signs the Informed Consent and Research Authorization document
5. Patient is able to read and speak English.

Exclusion Criteria:

1. Patient is under the age of 21
2. Patient's primary diagnosis is not osteoarthritis
3. Patient is unable to read and speak English
4. History of previous DVT/PE
5. History of stroke, CABG, or A fib
6. Current smoker

Ages: 21 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Overall Satisfaction | 1-year postoperatively
  Overall Satisfaction with TKA using a Likert scale
Pain VAS | preoperatively, 6 weeks (± 2 weeks), and 1-year postoperatively
  Level of knee pain (scale of zero to ten) using the Visual Analog Scale (VAS)
KOOS JR | preoperatively, 6 weeks (± 2 weeks), and 1-year postoperatively
  KOOS JR questionnaire
Forgotten Joint Score | preoperatively, 6 weeks (± 2 weeks), and 1-year postoperatively
  FJS-12 questionnaire
PROMIS-10 Mental and Physical Health scores | preoperatively and 1-year postoperatively
  PROMIS-10 Global Health questionnaire
Incidence of revision TKA | 1 year postop
  postoperative complication requiring a revision total knee arthroplasty
non-revision complication | 1 year postop
  postoperative complication requiring a non-revision procedure

SECONDARY OUTCOMES:
Active ROM | preoperatively, 6 weeks (± 2 weeks), and 1-year postoperatively
  Active knee range of motion: active extension, active flexion

CONTACTS AND LOCATIONS:
Locations (1):
- UofL Health, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Undecided